CLINICAL TRIAL: NCT05816369
Title: Taste and Smell Alterations and Oral Nutritional Supplement (ONS) Preferences in Patients With Cancer
Brief Title: Oral Nutritional Supplement Preferences in Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Smartfish AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Cancer Taste Study
Record Dates: First submitted 2023-03-15; First posted 2023-04-18 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Neoplasms; Malnutrition
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taste preferences of five ONS flavors (Experimental): Taste session with corresponding questionnaires
  Interventions: Other: Taste session of five ONS flavors

INTERVENTIONS:
Other: Taste session of five ONS flavors — Patients will taste a small sample (30 mL) of five ONS flavors and report their taste experiences by completing questionnaires of each flavor during the taste session. Participants will also complete a malnutrition risk screening (MST), a three-day food diary, questionnaires of self-reported taste and smell changes (TSS), and quality of life (RAND-36).

SUMMARY:
Patients diagnosed with cancer have a particularly high risk of developing malnutrition due to the disease itself and due to symptoms of cancer treatments that can affect food intake such as reduced appetite, nausea, fatigue, and alterations in taste and smell. Nutritional treatment is essential in the prevention and treatment of malnutrition. Oral nutritional supplements (ONS) are often recommended to cancer patients who need to increase their nutritional intake and are unable to meet their nutritional requirements by consumption of normal food alone. However, patient compliance with ONS depends on sensory acceptability of such products. Therefore, the objective of this study is to investigate preferences of sensory characteristics of ONS among cancer patients. Additionally, possible associations between taste and smell alterations and dietary intake, malnutrition risk, and quality of life will be investigated. The results from this study will optimize recommendations of ONS in the clinical setting and encourage new efforts among manufacturers in developing acceptable sensory characteristics of ONS to cancer patients. Findings from this study will contribute to improving nutritional treatment for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients diagnosed with lung cancer
* Patients receiving cancer treatment of different types
* Age 18 years or more
* Provided signed informed consent
* Understand written and oral Norwegian

Exclusion Criteria:

* Severe mental or cognitive disorders
* Contraindication to consume ONS (dysphagia, inability to swallow oral nutritional supplements)
* Allergic or intolerant to any of the ingredients in the ONS
* Terminally ill patients (<3 months to live)
* A clinically significant disease or condition that could, in the investigator's opinion make the patient unfit for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Flavor liking of five different oral nutritional supplement flavors. | 30 minutes
  To evaluate patient liking of five different oral nutritional supplement flavors using a taste test and a questionnaire with a 9-point Hedonic scale (possible score from 1 to 9) assessing flavor liking. A higher score indicates better liking.

SECONDARY OUTCOMES:
Self-reported taste and smell alterations. | 10 minutes
  Using the 16-item questionnaire Taste and Smell Survey (TSS). TSS consists of nine questions regarding changes in the sense of taste (possible score 0-10), five questions regarding changes in the sense of smell (possible score 0-6), and two global questions regarding quality of life. A higher total score indicates a higher number of aspects of taste and smell alterations.
Prevalence of malnutrition risk. | 5 minutes
  Malnutrition risk will be defined using the two-item questionnaire Malnutrition Screening Tool (MST). MST consists of one question regarding changes in weight (possible score 0-4) and one questions regarding changes in food intake (possible score 0-1). A total score of 2 or more defines a patient to be at risk of malnutrition.
Dietary intake. | 3 days
  Dietary intake will be defined using a three-day patient food diary. The three-day patient food diary consists of two reports from week days and one report from a weekend day. Patients will report everything that is consumed during these selected days.The average intake of macro- and micronutrients will be calculated.
Quality of life. | 10 minutes
  Using the 36-item questionnaire RAND-36. RAND-36 consists of eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions (possible score 0-100). A lower score indicates poorer quality of life.
Flavor liking with and without the presence of taste and smell alterations by the 16-item questionnaire Taste and Smell Survey (TSS). | 30 minutes
  Using a 9-point Hedonic scale (possible score from 1 to 9) assessing flavor liking. A higher score indicates better liking. The presence of self reported taste and smell alterations will be defined by the answer response "yes" to any of the six questions in the Taste and Smell Survey (TSS) addressing the presence of taste and smell alterations.
Liking of ONS characteristics with and without the presence of taste and smell alterations by the 16-item questionnaire Taste and Smell Survey (TSS). | 30 minutes
  Using a taste test and questionnaires with a 5-point Just About Right (JAR) scale regarding flavor intensity, acidity, sweetness, and viscosity. The presence of self reported taste and smell alterations will be defined by the answer response "yes" to any of the six questions in the Taste and Smell Survey (TSS) addressing the presence of taste and smell alterations.

CONTACTS AND LOCATIONS:
Overall Officials: Simon N Dankel, Professor, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No